CLINICAL TRIAL: NCT00582114
Title: Hypertension in Hemodialysis Patients
Brief Title: Hypertension in Hemodialysis Patients (Aim 3)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped by data safety monitoring board
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0306-13; R01DK062030 (NIH); NIH-NIDDK-5RO1-062030
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-12

CONDITIONS: Hemodialysis; Hypertension; Left Ventricular Hypertrophy
Keywords: Hemodialysis; Hypertension; Left ventricular hypertrophy
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — Lisinopril; Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Atenolol
  Interventions: Drug: Atenolol
- 2 (Experimental): Lisinopril
  Interventions: Drug: Lisinopril

INTERVENTIONS:
Drug: Lisinopril — Patients will be randomized into two groups, one that is beta blocker based, the other angiotensin converting enzyme (ACE) inhibitor (lisinopril) based. Patients who are on no medications will receive atenolol 25 mg. t.i.w. or lisinopril 10 mg. t.i.w. for one month at the end of which, dose will be titrated to twice the drug doses following monthly interval to another doubling of dose. If BP is still poorly controlled felodipine will be added. Other antihypertensive therapies will be added to control home BP to <140/90 mm Hg.
  Arms: 2
Drug: Atenolol — Patients will be randomized into two groups, one that is beta blocker based, the other angiotensin converting enzyme (ACE) inhibitor (lisinopril) based. Patients who are on no medications will receive atenolol 25 mg. t.i.w. or lisinopril 10 mg. t.i.w. for one month at the end of which, dose will be titrated to twice the drug doses following monthly interval to another doubling of dose. If BP is still poorly controlled felodipine will be added. Other antihypertensive therapies will be added to control home BP to <140/90 mm Hg.
  Arms: 1

SUMMARY:
We will directly test the hypothesis that an initial strategy of lisinopril-based therapy will be more effective than atenolol-based therapy in causing regression of left ventricular hypertrophy (LVH) over one year in patients with hemodialysis hypertension despite similar degree of BP reduction.

DETAILED DESCRIPTION:
This is a parallel group, active control, single-center, open-label, randomized controlled trial comparing the safety and efficacy of initial therapy with an angiotensin converting enzyme (ACE) inhibitor (lisinopril) vs. beta-blocker therapy (atenolol) each administered three times weekly after dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients on chronic hemodialysis for > 3 mos.
2. Compliance with hemodialysis treatments as defined by less than one missed dialysis per month
3. Hypertension as diagnosed by ambulatory blood pressure monitoring (ABPM) >135/75 mm Hg after participation in the ultrafiltration (UF) Trial, or those on no antihypertensive medications but unwilling to do UF Trial.
4. Presence of LVH on echocardiogram defined as left ventricular mass index (LVMi) >104 g/m2 in women and >116 g/m2 in men.
5. Willingness to give informed consent.

Exclusion criteria:

1. Vascular event (stroke, myocardial infarction or limb ischemia requiring bypass) within previous six months
2. Noncompliance with hemodialysis treatments
3. Known drug abuse
4. Chronic obstructive pulmonary disorder (COPD) requiring home oxygen
5. Congestive Heart Failure Class III or IV.
6. Body mass index > 40 kg/m2.
7. Known contraindication to atenolol (severe heart failure, bradycardia, bronchial asthma, intolerance or allergy) or lisinopril (cough, pregnancy, intolerance or allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Agarwal, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Agarwal R, Sinha AD, Pappas MK, Abraham TN, Tegegne GG. Hypertension in hemodialysis patients treated with atenolol or lisinopril: a randomized controlled trial. Nephrol Dial Transplant. 2014 Mar;29(3):672-81. doi: 10.1093/ndt/gft515. Epub 2014 Jan 6. PMID 24398888

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisinopril: Lisinopril: Patients will be randomized into two groups, one that is beta blocker based, the other ACE inhibitor (lisinopril) based. Patients who are on no medications will receive atenolol 25 mg. t.i.w. or lisinopril 10 mg. t.i.w. for one month at the end of which, dose will be titrated to twice the drug doses following monthly interval to another doubling of dose. If BP is still poorly controlled felodipine will be added. Other antihypertensive therapies will be added to control home BP to <140/90 mm Hg.
Period: Overall Study
Arm/Group | Atenolol | Lisinopril
Started | 100 | 100
Completed | 58 | 46
Not Completed | 42 | 54
Not completed — Death | 4 | 4
Not completed — Kidney Transplant | 3 | 1
Not completed — Lost to Follow-up | 7 | 6
Not completed — Withdrawal by Subject | 8 | 16
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 0 | 6
Not completed — Stopped by data safety monitoring board | 19 | 20

BASELINE CHARACTERISTICS:
Groups:
- Atenolol: Atenolol: Patients will be randomized into two groups, one that is beta blocker based, the other ACE inhibitor (lisinopril) based. Patients who are on no medications will receive atenolol 25 mg. t.i.w. or lisinopril 10 mg. t.i.w. for one month at the end of which, dose will be titrated to twice the drug doses following monthly interval to another doubling of dose. If BP is still poorly controlled felodipine will be added. Other antihypertensive therapies will be added to control home BP to <140/90 mm Hg.
- Total: Total of all reporting groups
Arm/Group | Atenolol | Lisinopril | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (11.7) | 53.1 (13.5) | 52.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 42 | 69
  Male | 73 | 58 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 99 | 100 | 199
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Blacks | 86 | 86 | 172
  Non-blacks | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200
Etiology of chronic kidney disease [Number; unit: participants]
  Diabetes mellitus | 29 | 27 | 56
  Hypertension | 54 | 46 | 100
  Glomerulonephritis | 4 | 5 | 9
  Polycystic kidney disease | 0 | 1 | 1
  Other etiologies | 13 | 21 | 34
Dialysis vintage [Mean (Standard Deviation); unit: years] | 4.2 (4.4) | 3.9 (4.2) | 4.1 (4.3)
Anuric [Number; unit: participants] | 68 | 66 | 134
Education [Mean (Standard Deviation); unit: years] | 12 (2) | 12 (2) | 12 (2)
Comorbid conditions [Number; unit: participants]
  Diabetes mellitus | 43 | 43 | 86
  Hospitalized heart failure | 25 | 37 | 62
  Coronary artery disease | 22 | 31 | 53
  Coronary revascularization | 4 | 15 | 19
  Cerebrovascular disease | 13 | 20 | 33
  Peripheral vascular disease | 10 | 11 | 21
Marital status [Number; unit: participants]
  Single | 53 | 56 | 109
  Married | 23 | 19 | 42
  Divorced/separated | 18 | 15 | 33
  Widowed | 6 | 10 | 16
Employed [Number; unit: participants]
  Working | 11 | 7 | 18
  Not working | 67 | 70 | 137
  Retired | 22 | 23 | 45
Income [Number; unit: participants]
  < $25,000 | 84 | 80 | 164
  >= $25,000 | 10 | 7 | 17
  Refused | 6 | 13 | 19
Smoking [Number; unit: participants]
  Current smoker | 43 | 43 | 86
  Non-smoker | 57 | 57 | 114
Alcohol [Number; unit: participants]
  Drinks alcohol | 27 | 19 | 46
  Does not drink alcohol | 73 | 81 | 154
Height [Mean (Standard Deviation); unit: inches] | 68.3 (4.1) | 67.6 (3.7) | 67.9 (3.9)
Weight [Mean (Standard Deviation); unit: kg] | 85.1 (21.7) | 80.9 (24.3) | 83 (23.1)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (7) | 27.5 (8.3) | 27.9 (7.7)
Access type [Number; unit: participants]
  Fistula | 59 | 59 | 118
  Graft | 16 | 14 | 30
  Catheter | 25 | 27 | 52
Blood flow rate [Mean (Standard Deviation); unit: mL/min] | 394.3 (30.9) | 392.4 (36.4) | 393.4 (33.7)
Dialysate flow rate [Mean (Standard Deviation); unit: mL/min] | 779.6 (61.9) | 761.3 (82) | 770.4 (73)
Dialysis duration [Mean (Standard Deviation); unit: minutes]
  Prescribed dialysis duration | 239.4 (19) | 239.4 (25.9) | 239.4 (22.7)
  Delivered dialysis duration | 224.1 (34.7) | 219.8 (33.7) | 222 (34.2)
Urea reduction ratio [Mean (Standard Deviation); unit: %] | 74 (8) | 76 (8) | 75 (8)
Albumin [Mean (Standard Deviation); unit: g/dL] | 3.6 (0.5) | 3.6 (0.5) | 3.6 (0.5)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 11.3 (1.2) | 11.3 (1.4) | 11.3 (1.3)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 10.3 (3.5) | 10 (3.6) | 10.1 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: The Primary End Point is the Regression of Left Ventricular Hypertrophy (LVH) by Echocardiographic Criteria From Baseline to 1 Year.
Description: The primary outcome of the study was the average reduction in left ventricular mass indexed for body surface area from baseline to 1 year. A mixed model was used with left ventricular mass index (LVMI) as the outcome variable. Fixed effects were indicator variables for time, treatment and their interaction. Random effect was subject and statistical inference was made using the maximum likelihood estimator. No imputation was made for missing data.
Time Frame: Baseline, 6 months, 12 months
Population: The primary outcome of the study was the average reduction in left ventricular mass indexed for body surface area from baseline to 1 year. The analysis was performed by intention to treat, if the patient received at least one dose of the randomized drug regardless of the availability of a post-baseline echocardiogram.
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Atenolol | Lisinopril
Number analyzed (Participants) | 100 | 100
g/m^2
  LVMI Change from baseline, 6 months | -8.4 (5.1) | -3.4 (5.5)
  LVMI Change from baseline, 12 months | -21.5 (5.7) | -15.1 (6.2)

2. Other Pre Specified Outcome: Serious Adverse Events and Cardiovascular Events That Led to Trial Termination
Description: Cardiovascular events were counted by subject and included the following: myocardial infarction (MI), stroke, hospitalization for congestive heart failure (CHF), hospitalized angina, arrhythmias, cardiac arrest, coronary revascularization and heart valve replacement. Adverse events reported are those during the course of 12 months of participation in the trial. All serious adverse events were adjudicated by R.A. and A.D.S. who were masked to the drug assignment at the time of adjudication. The duration of participation in the study per subject, which according to the trial design could be up to 12 months, was determined. The cardiovascular event rate was calculated by treatment group assignment. Incidence rate ratio (IRR) by treatment was then determined along with the 95% confidence intervals (95% CIs). As a post hoc analysis, we also determined the narrower definition of cardiovascular events per group that included MI, stroke, CHF, or cardiovascular death.
Time Frame: 1 yr
Measure: Number; unit: events/100 patient-years
Arm/Group | Atenolol | Lisinopril
Number analyzed (Participants) | 100 | 100
events/100 patient-years
  Incidence rate, cardiovasular events | 24.6 | 58
  Incidence rate, combined MI, stroke, CHF, CV death | 13.5 | 31
  Incidence rate, congest heart failure | 6.2 | 20.2
  Incidence rate, all-cause hospitalizations | 89.9 | 144.3
Statistical Analysis 1: Comparison: Atenolol vs Lisinopril; Cardiovascular events were counted by subject and included the following: myocardial infarction, stroke, hospitalization for congestive heart failure, hospitalized angina, arrhythmias, cardiac arrest, coronary revascularization and heart valve replacement. The duration of participation in the study per subject, which according to the trial design could be up to 12 months, was determined. Incidence rate ratio (IRR) by treatment was then determined along with the 95%confidence intervals (95% CIs); Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Hazard Ratio (HR) = 2.36, 95% CI 2-sided [1.36 to 4.23]
Statistical Analysis 2: Comparison: Atenolol vs Lisinopril; As a post hoc analysis, we determined the narrower definition of cardiovascular events per group that included myocardial infarction, stroke, congestive heart failure or cardiovascular death. The duration of participation in the study per subject, which according to the trial design could be up to 12 months, was determined. Incidence rate ratio (IRR) by treatment was then determined along with the 95%confidence intervals (95% CIs); Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Hazard Ratio (HR) = 2.29, 95% CI 2-sided [1.07 to 5.21]
Statistical Analysis 3: Comparison: Atenolol vs Lisinopril; Hospitalization for congestive heart failure between groups was analyzed. The duration of participation in the study per subject, which according to the trial design could be up to 12 months, was determined. Incidence rate ratio (IRR) by treatment was then determined along with the 95%confidence intervals; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Hazard Ratio (HR) = 3.13, 95% CI 2-sided [1.08 to 10.99]
Statistical Analysis 4: Comparison: Atenolol vs Lisinopril; All-cause hospitalizations between groups were analyzed. The duration of participation in the study per subject, which according to the trial design could be up to 12 months, was determined. Incidence rate ratio (IRR) by treatment was then determined along with the 95%confidence intervals; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Hazard Ratio (HR) = 1.61, 95% CI 2-sided [1.18 to 2.19]

ADVERSE EVENTS:
Arm/Group | Atenolol | Lisinopril
Serious Adverse Events (participants affected / at risk) | 58/100 | 70/100
Other Adverse Events (participants affected / at risk) | 44/100 | 29/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atenolol (N=100) | Lisinopril (N=100)
Infections (Infections and infestations) | 24 (30) | 20 (29)
Access-related (Renal and urinary disorders) | 17 (24) | 19 (30)
Central nervous system (Nervous system disorders) | 3 (3) | 3 (5)
Cancer-related complications (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 2 (3)
Angina (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 2 (2) | 3 (5)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Congestive heart failure (Cardiac disorders) | 5 (5) | 10 (15)
Myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3)
Peripheral vascular disease (Cardiac disorders) | 1 (1) | 5 (6)
Revascularization (Cardiac disorders) | 3 (4) | 4 (4)
Stroke (Cardiac disorders) | 2 (2) | 2 (2)
Valve replacement surgery (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular death (Cardiac disorders) | 2 (2) | 3 (3)
Noncardiovascular death (General disorders) | 2 (2) | 1 (1)
Fractures (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Parathyroidectomy (Endocrine disorders) | 3 (3) | 1 (1)
Biliary-related (Hepatobiliary disorders) | 1 (1) | 2 (2)
Bowel-related (Gastrointestinal disorders) | 3 (3) | 5 (5)
Falls (General disorders) | 6 (6) | 3 (3)
Gastrointestinal bleed (Gastrointestinal disorders) | 2 (4) | 5 (7)
Hypertensive crisis (General disorders) | 3 (3) | 10 (11)
Hyperglycemia (Endocrine disorders) | 1 (2) | 3 (3)
Hyperkalemia (Renal and urinary disorders) | 3 (3) | 10 (10)
Hypoglycemia (Endocrine disorders) | 2 (3) | 4 (4)
Hypotension with hospitalization (General disorders) | 6 (8) | 5 (5)
Miscellaneous (General disorders) | 12 (14) | 18 (24)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atenolol (N=100) | Lisinopril (N=100)
Fatigue (General disorders) | 20 (25) | 6 (12)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (6) | 6 (6)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (4)
bradycardia (General disorders) | 2 (3) | 1 (1)
Intradialytic hypotension (General disorders) | 6 (7) | 4 (4)
tachycardia (General disorders) | 1 (1) | 1 (1)
Dialysis access-related events (General disorders) | 0 (0) | 1 (1)
Hypertension (General disorders) | 1 (1) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Other (General disorders) | 19 (23) | 17 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No